CLINICAL TRIAL: NCT01753245
Title: CARDIOVASCULAR RISK FACTORS IN A SPANISH POPULATION OF PATIENTS WITH MODERATE-TO-SEVERE PSORIASIS VULGARIS, WITH OR WITHOUT ARTHRITIS, TREATED WITH ANTI-TNF IN REAL CLINICAL PRACTICE. ANALYSIS OF THE INFLUENCE OF METABOLIC SYNDROME ON TREATMENT EFFICACY.
Brief Title: Analysis Of The Influence Of Metabolic Syndrome On Treatment Efficacy With Anti-Tnf In Moderate-Severe Psoriasis In Real Clinical Practice.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Juan Ruano (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Juan Ruano, M.D., Ph.D., Ms.C., Hospital Universitario Reina Sofia de Cordoba
Organization: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Other Study IDs: JRR-ANT-2012-01; JRR-ANT-2012-01 (Other: Agencia Española de Medicamentos y Productos Sanitarios)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Psoriasis Vulgaris; Metabolic Syndrome
Keywords: Anti-TNF drugs efficacy; Moderate-to-severe psoriasis vulgaris; Gene polymorphism
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-Metabolic Syndrome: Patients without Metabolic Syndrome criteria (OMS).
- Metabolic Syndrome: Patients with Metabolic Syndrome criteria (OMS).

SUMMARY:
It has been reported in various epidemiological studies that patients with moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, have an increased frequency of cardiovascular risk factors, such as hypertension, obesity, type-2 diabetes mellitus (T2DM, and metabolic syndrome (MetS). The presence of endothelial dysfunction in early stages, especially in moderate-to-severe plaque psoriasis forms, could explain the higher prevalence of cardiovascular disease and mortality observed in this population. Existing evidence showing improvement in psoriasis after correcting some factors, such as obesity or hypercholesterolemia, and the reduction of certain surrogate markers of cardiovascular risk with different modalities of psoriasis treatment suggest a biological interaction between the two diseases beyond mere epidemiological association. Recently published results support this hypothesis and suggest that the link between psoriasis and cardiovascular disease could be the existence of an inflammatory state in different organs, including skin, joints, adipose and hepatic tissue, and vascular endothelium (16). Patients with MetS have an increased risk of developing T2DM and cardiovascular disease. This syndrome is characterized by the association of an adipose tissue inflammatory state and diminished sensitivity to insulin. In recent years, a new mechanism participating in the development of MetS has been added: the Wnt signaling pathway. Polymorphisms in genes of the Wnt signaling pathway have been associated with metabolic abnormalities that predispose to cardiovascular disease, the development of moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, and response to treatment with anti-TNF-alpha.

This study aims to describe the cardiovascular risk factors of a Spanish population of patients with moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis,treated with anti-TNF under routine clinical practice conditions. Possible differences in efficacy relative to the presence or absence of criteria of metabolic syndrome will be analyzed. Similarly, we will explore the role of markers of inflammatory activity and genetic polymorphisms in the Wnt pathway in predicting response to treatment during the first year.

DETAILED DESCRIPTION:
1. Eligibility criteria:

   1.1. Inclusion criteria:
   1. -Age >18 ys.
   2. -Male and female.
   3. -Moderate-to-severe psoriasis vulgaris, with or without psoriatic arthritis.
   4. -Treated with anti-TNF drugs (infliximab, etanercept, adalimumab). 1.2. Exclusion criteria:

   <!-- -->

   1. -Enrolled in another clinical trial.
   2. -Lack of clinical information at the hospital database.
2. Objectives:

2.1. Primary objective: Evaluate the efficacy of anti-TNF- drugs in the treatment of patients with moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, in terms of the presence or absence of cardiovascular risk factors, including metabolic syndrome.

2.2. Secondary objectives:

* 2.2.1. Analyze the possible modulatory role of genetic factors, such as Wnt pathway's gene polymorphisms, and other nongenetic factors on responsiveness to treatment with anti-TNF drugs in the overall study population and in the subgroup of patients with metabolic syndrome.
* 2.2.2. Describe the cardiovascular risk factors in patients with moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, treated with anti-TNF- in the Spanish population under routine clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe psoriasis treated >1 ys with anti-TNFalpha drugs
* Age >18 ys/<80 ys
* With or without psoriatic arthritis

Exclusion Criteria:

* Enrolled in another trial
* Lack of clinical information
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Moderate-to-severe psoriasis treated >1 ys with anti-TNFalpha drugs at Reina Sofia University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Role of Metabolic Syndrome on anti-TNF-drug efficacy. | After one year of treatment
  Evaluate the efficacy of anti-TNF-drugs in themoderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, in terms of the presence or absence of cardiovascular risk factors, including metabolic syndrome.

SECONDARY OUTCOMES:
Effect of 'Wnt pathway' genetic polymorphisms on anti-TNF-drug efficacy | First year of treament
  Analyze the possible modulatory role of genetic factors, such as Wnt polymorphisms, and nongenetic factors on responsiveness to treatment with anti-TNF drugs in the overall study population and in the subgroup of patients with metabolic syndrome.

OTHER OUTCOMES:
Cardiovascular disease factors | First year of treatment
  Describe the cardiovascular risk factors in patients with moderate-to-severe plaque psoriasis, with or without associated psoriatic arthritis, treated with anti-TNF- in the Spanish population under routine clinical practice conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ruano, M.D., Ph.D., Ms. C., Principal Investigator — Departament of Dermatology. Reina Sofia University Hospital.
Locations (1):
- Department of Dermatology. Reina Sofia University Hospital., Córdoba, Cordoba, Spain

REFERENCES:
- [Background] Gisondi P, Farina S, Giordano MV, Girolomoni G. Usefulness of the framingham risk score in patients with chronic psoriasis. Am J Cardiol. 2010 Dec 15;106(12):1754-7. doi: 10.1016/j.amjcard.2010.08.016. Epub 2010 Nov 4. PMID 21055711
- [Background] Choi WJ, Park EJ, Kwon IH, Kim KH, Kim KJ. Association between Psoriasis and Cardiovascular Risk Factors in Korean Patients. Ann Dermatol. 2010 Aug;22(3):300-6. doi: 10.5021/ad.2010.22.3.300. Epub 2010 Aug 5. PMID 20711266
- [Background] Limbrock GJ, Hoyer H, Scheying H. Drooling, chewing and swallowing dysfunctions in children with cerebral palsy: treatment according to Castillo-Morales. ASDC J Dent Child. 1990 Nov-Dec;57(6):445-51. PMID 2147927
- [Background] Karadag AS, Yavuz B, Ertugrul DT, Akin KO, Yalcin AA, Deveci OS, Ata N, Kucukazman M, Dal K. Is psoriasis a pre-atherosclerotic disease? Increased insulin resistance and impaired endothelial function in patients with psoriasis. Int J Dermatol. 2010 Jun;49(6):642-6. doi: 10.1111/j.1365-4632.2009.04358.x. PMID 20618468
- [Background] Prey S, Paul C, Bronsard V, Puzenat E, Gourraud PA, Aractingi S, Aubin F, Bagot M, Cribier B, Joly P, Jullien D, Le Maitre M, Richard-Lallemand MA, Ortonne JP. Cardiovascular risk factors in patients with plaque psoriasis: a systematic review of epidemiological studies. J Eur Acad Dermatol Venereol. 2010 Apr;24 Suppl 2:23-30. doi: 10.1111/j.1468-3083.2009.03564.x. PMID 20443997
- [Background] Zindanci I, Albayrak O, Kavala M, Kocaturk E, Can B, Sudogan S, Koc M. Prevalence of metabolic syndrome in patients with psoriasis. ScientificWorldJournal. 2012;2012:312463. doi: 10.1100/2012/312463. Epub 2012 Apr 24. PMID 22654590
- [Background] Alsufyani MA, Golant AK, Lebwohl M. Psoriasis and the metabolic syndrome. Dermatol Ther. 2010 Mar-Apr;23(2):137-43. doi: 10.1111/j.1529-8019.2010.01307.x. PMID 20415820
- [Background] Martyn-Simmons CL, Ranawaka RR, Chowienczyk P, Crook MA, Marber MS, Smith CH, Barker JN. A prospective case-controlled cohort study of endothelial function in patients with moderate to severe psoriasis. Br J Dermatol. 2011 Jan;164(1):26-32. doi: 10.1111/j.1365-2133.2010.10031.x. Epub 2010 Nov 8. PMID 20819085
- [Background] Ardic I, Kaya MG, Yarlioglues M, Karadag Z, Dogan A, Yildiz H, Dogdu O, Zencir C, Aktas E, Ergin A. Impaired aortic elastic properties in normotensive patients with psoriasis. Blood Press. 2010 Dec;19(6):351-8. doi: 10.3109/08037051.2010.505322. Epub 2010 Jul 16. PMID 20635857
- [Background] Abuabara K, Azfar RS, Shin DB, Neimann AL, Troxel AB, Gelfand JM. Cause-specific mortality in patients with severe psoriasis: a population-based cohort study in the U.K. Br J Dermatol. 2010 Sep;163(3):586-92. doi: 10.1111/j.1365-2133.2010.09941.x. PMID 20633008
- [Background] Gisondi P, Del Giglio M, Di Francesco V, Zamboni M, Girolomoni G. Weight loss improves the response of obese patients with moderate-to-severe chronic plaque psoriasis to low-dose cyclosporine therapy: a randomized, controlled, investigator-blinded clinical trial. Am J Clin Nutr. 2008 Nov;88(5):1242-7. doi: 10.3945/ajcn.2008.26427. PMID 18996858
- [Background] Ghazizadeh R, Tosa M, Ghazizadeh M. Clinical improvement in psoriasis with treatment of associated hyperlipidemia. Am J Med Sci. 2011 May;341(5):394-8. doi: 10.1097/MAJ.0b013e3181ff8eeb. PMID 21233693
- [Background] Boehncke S, Salgo R, Garbaraviciene J, Beschmann H, Hardt K, Diehl S, Fichtlscherer S, Thaci D, Boehncke WH. Effective continuous systemic therapy of severe plaque-type psoriasis is accompanied by amelioration of biomarkers of cardiovascular risk: results of a prospective longitudinal observational study. J Eur Acad Dermatol Venereol. 2011 Oct;25(10):1187-93. doi: 10.1111/j.1468-3083.2010.03947.x. Epub 2011 Jan 17. PMID 21241371
- [Background] Mehta NN, Yu Y, Saboury B, Foroughi N, Krishnamoorthy P, Raper A, Baer A, Antigua J, Van Voorhees AS, Torigian DA, Alavi A, Gelfand JM. Systemic and vascular inflammation in patients with moderate to severe psoriasis as measured by [18F]-fluorodeoxyglucose positron emission tomography-computed tomography (FDG-PET/CT): a pilot study. Arch Dermatol. 2011 Sep;147(9):1031-9. doi: 10.1001/archdermatol.2011.119. Epub 2011 May 16. PMID 21576552
- [Background] Bissonnette R, Tardif JC, Harel F, Pressacco J, Bolduc C, Guertin MC. Effects of the tumor necrosis factor-alpha antagonist adalimumab on arterial inflammation assessed by positron emission tomography in patients with psoriasis: results of a randomized controlled trial. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):83-90. doi: 10.1161/CIRCIMAGING.112.975730. Epub 2012 Nov 30. PMID 23204039
- [Background] Lusis AJ, Attie AD, Reue K. Metabolic syndrome: from epidemiology to systems biology. Nat Rev Genet. 2008 Nov;9(11):819-30. doi: 10.1038/nrg2468. PMID 18852695
- [Background] Smolich BD, McMahon JA, McMahon AP, Papkoff J. Wnt family proteins are secreted and associated with the cell surface. Mol Biol Cell. 1993 Dec;4(12):1267-75. doi: 10.1091/mbc.4.12.1267. PMID 8167409
- [Background] Sethi JK, Vidal-Puig A. Wnt signalling and the control of cellular metabolism. Biochem J. 2010 Mar 15;427(1):1-17. doi: 10.1042/BJ20091866. PMID 20226003
- [Background] George SJ. Wnt pathway: a new role in regulation of inflammation. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):400-2. doi: 10.1161/ATVBAHA.107.160952. No abstract available. PMID 18296599
- [Background] Bilkovski R, Schulte DM, Oberhauser F, Mauer J, Hampel B, Gutschow C, Krone W, Laudes M. Adipose tissue macrophages inhibit adipogenesis of mesenchymal precursor cells via wnt-5a in humans. Int J Obes (Lond). 2011 Nov;35(11):1450-4. doi: 10.1038/ijo.2011.6. Epub 2011 Feb 1. PMID 21285942
- [Background] Ouchi N, Higuchi A, Ohashi K, Oshima Y, Gokce N, Shibata R, Akasaki Y, Shimono A, Walsh K. Sfrp5 is an anti-inflammatory adipokine that modulates metabolic dysfunction in obesity. Science. 2010 Jul 23;329(5990):454-7. doi: 10.1126/science.1188280. Epub 2010 Jun 17. PMID 20558665
- [Background] Isakson P, Hammarstedt A, Gustafson B, Smith U. Impaired preadipocyte differentiation in human abdominal obesity: role of Wnt, tumor necrosis factor-alpha, and inflammation. Diabetes. 2009 Jul;58(7):1550-7. doi: 10.2337/db08-1770. Epub 2009 Apr 7. PMID 19351711
- [Background] Salpea KD, Gable DR, Cooper JA, Stephens JW, Hurel SJ, Ireland HA, Feher MD, Godsland IF, Humphries SE. The effect of WNT5B IVS3C>G on the susceptibility to type 2 diabetes in UK Caucasian subjects. Nutr Metab Cardiovasc Dis. 2009 Feb;19(2):140-5. doi: 10.1016/j.numecd.2008.02.009. Epub 2008 Jun 13. PMID 18555673
- [Background] Kim IC, Cha MH, Kim DM, Lee H, Moon JS, Choi SM, Kim KS, Yoon Y. A functional promoter polymorphism -607G>C of WNT10B is associated with abdominal fat in Korean female subjects. J Nutr Biochem. 2011 Mar;22(3):252-8. doi: 10.1016/j.jnutbio.2010.02.002. Epub 2010 Jun 25. PMID 20579865
- [Background] Haupt A, Thamer C, Heni M, Ketterer C, Machann J, Schick F, Machicao F, Stefan N, Claussen CD, Haring HU, Fritsche A, Staiger H. Gene variants of TCF7L2 influence weight loss and body composition during lifestyle intervention in a population at risk for type 2 diabetes. Diabetes. 2010 Mar;59(3):747-50. doi: 10.2337/db09-1050. Epub 2009 Dec 22. PMID 20028944
- [Background] Delgado-Lista J, Perez-Martinez P, Garcia-Rios A, Phillips CM, Williams CM, Gulseth HL, Helal O, Blaak EE, Kiec-Wilk B, Basu S, Drevon CA, Defoort C, Saris WH, Wybranska I, Riserus U, Lovegrove JA, Roche HM, Lopez-Miranda J. Pleiotropic effects of TCF7L2 gene variants and its modulation in the metabolic syndrome: from the LIPGENE study. Atherosclerosis. 2011 Jan;214(1):110-6. doi: 10.1016/j.atherosclerosis.2010.10.027. Epub 2010 Nov 3. PMID 21115178
- [Background] Phillips CM, Goumidi L, Bertrais S, Field MR, McManus R, Hercberg S, Lairon D, Planells R, Roche HM. Dietary saturated fat, gender and genetic variation at the TCF7L2 locus predict the development of metabolic syndrome. J Nutr Biochem. 2012 Mar;23(3):239-44. doi: 10.1016/j.jnutbio.2010.11.020. Epub 2011 May 2. PMID 21543200
- [Background] Liu PH, Chang YC, Jiang YD, Chen WJ, Chang TJ, Kuo SS, Lee KC, Hsiao PC, Chiu KC, Chuang LM. Genetic variants of TCF7L2 are associated with insulin resistance and related metabolic phenotypes in Taiwanese adolescents and Caucasian young adults. J Clin Endocrinol Metab. 2009 Sep;94(9):3575-82. doi: 10.1210/jc.2009-0609. Epub 2009 Jun 9. PMID 19509102
- [Background] Muendlein A, Saely CH, Geller-Rhomberg S, Sonderegger G, Rein P, Winder T, Beer S, Vonbank A, Drexel H. Single nucleotide polymorphisms of TCF7L2 are linked to diabetic coronary atherosclerosis. PLoS One. 2011 Mar 15;6(3):e17978. doi: 10.1371/journal.pone.0017978. PMID 21423583
- [Background] Guo YF, Xiong DH, Shen H, Zhao LJ, Xiao P, Guo Y, Wang W, Yang TL, Recker RR, Deng HW. Polymorphisms of the low-density lipoprotein receptor-related protein 5 (LRP5) gene are associated with obesity phenotypes in a large family-based association study. J Med Genet. 2006 Oct;43(10):798-803. doi: 10.1136/jmg.2006.041715. Epub 2006 May 24. PMID 16723389
- [Background] Saarinen A, Saukkonen T, Kivela T, Lahtinen U, Laine C, Somer M, Toiviainen-Salo S, Cole WG, Lehesjoki AE, Makitie O. Low density lipoprotein receptor-related protein 5 (LRP5) mutations and osteoporosis, impaired glucose metabolism and hypercholesterolaemia. Clin Endocrinol (Oxf). 2010 Apr;72(4):481-8. doi: 10.1111/j.1365-2265.2009.03680.x. Epub 2009 Aug 5. PMID 19673927
- [Background] Sarzani R, Salvi F, Bordicchia M, Guerra F, Battistoni I, Pagliariccio G, Carbonari L, Dessi-Fulgheri P, Rappelli A. Carotid artery atherosclerosis in hypertensive patients with a functional LDL receptor-related protein 6 gene variant. Nutr Metab Cardiovasc Dis. 2011 Feb;21(2):150-6. doi: 10.1016/j.numecd.2009.08.004. Epub 2009 Oct 14. PMID 19833493
- [Background] Tomaszewski M, Charchar FJ, Barnes T, Gawron-Kiszka M, Sedkowska A, Podolecka E, Kowalczyk J, Rathbone W, Kalarus Z, Grzeszczak W, Goodall AH, Samani NJ, Zukowska-Szczechowska E. A common variant in low-density lipoprotein receptor-related protein 6 gene (LRP6) is associated with LDL-cholesterol. Arterioscler Thromb Vasc Biol. 2009 Sep;29(9):1316-21. doi: 10.1161/ATVBAHA.109.185355. Epub 2009 Aug 10. PMID 19667113
- [Background] Liu YJ, Liu XG, Wang L, Dina C, Yan H, Liu JF, Levy S, Papasian CJ, Drees BM, Hamilton JJ, Meyre D, Delplanque J, Pei YF, Zhang L, Recker RR, Froguel P, Deng HW. Genome-wide association scans identified CTNNBL1 as a novel gene for obesity. Hum Mol Genet. 2008 Jun 15;17(12):1803-13. doi: 10.1093/hmg/ddn072. Epub 2008 Mar 5. PMID 18325910
- [Background] Morikawa T, Kuchiba A, Yamauchi M, Meyerhardt JA, Shima K, Nosho K, Chan AT, Giovannucci E, Fuchs CS, Ogino S. Association of CTNNB1 (beta-catenin) alterations, body mass index, and physical activity with survival in patients with colorectal cancer. JAMA. 2011 Apr 27;305(16):1685-94. doi: 10.1001/jama.2011.513. PMID 21521850
- [Background] Reischl J, Schwenke S, Beekman JM, Mrowietz U, Sturzebecher S, Heubach JF. Increased expression of Wnt5a in psoriatic plaques. J Invest Dermatol. 2007 Jan;127(1):163-9. doi: 10.1038/sj.jid.5700488. Epub 2006 Jul 20. PMID 16858420
- [Background] Gudjonsson JE, Johnston A, Stoll SW, Riblett MB, Xing X, Kochkodan JJ, Ding J, Nair RP, Aphale A, Voorhees JJ, Elder JT. Evidence for altered Wnt signaling in psoriatic skin. J Invest Dermatol. 2010 Jul;130(7):1849-59. doi: 10.1038/jid.2010.67. Epub 2010 Apr 8. PMID 20376066
- [Background] Romanowska M, Evans A, Kellock D, Bray SE, McLean K, Donandt S, Foerster J. Wnt5a exhibits layer-specific expression in adult skin, is upregulated in psoriasis, and synergizes with type 1 interferon. PLoS One. 2009;4(4):e5354. doi: 10.1371/journal.pone.0005354. Epub 2009 Apr 28. PMID 19399181
- [Background] Suarez-Farinas M, Fuentes-Duculan J, Lowes MA, Krueger JG. Resolved psoriasis lesions retain expression of a subset of disease-related genes. J Invest Dermatol. 2011 Feb;131(2):391-400. doi: 10.1038/jid.2010.280. Epub 2010 Sep 23. PMID 20861854
- See also: Reina Sofia University Hospital — http://www.juntadeandalucia.es/servicioandaluzdesalud/hrs3